CLINICAL TRIAL: NCT06612112
Title: Investigation of the Relationship Between Trunk Balance and Trunk Position Sense, Wheelchair Skills and Functional Independence in Individuals With Thoracic Spinal Cord Injury
Brief Title: Trunk Balance and Functional Independence in Individuals With SCI
Acronym: SCI
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Yunus Emre Kundakçı, Associate Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2024/2-25
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-09

CONDITIONS: Spinal Cord Injury (SCI)
Keywords: Balance; Functional Independence; Trunk Position Sense; Spinal Cord Injury; Wheelchair Ability
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Thoracic SCI individuals: According to the ASIA (American Spinal Injury Association) Scale criteria, ASIA A patients had a complete lesion; ASIA B, ASIA C and ASIA D patients had an incomplete lesion.
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — No Interventions

SUMMARY:
This study investigates the relationship between trunk balance, position sense, wheelchair skills, and functional independence in individuals with thoracic spinal cord injury. It aims to understand how these factors interact and influence daily activities and overall quality of life.

DETAILED DESCRIPTION:
Sitting balance and wheelchair transfer activities are crucial for non-ambulatory spinal cord injury (SCI) patients to be able to perform activities of daily living. In addition, a comprehensive assessment of trunk balance is recommended in the literature to predict the risk of falls in these patients and to determine their functional independence. However, no study was found in the literature that included only patients with thoracic level involvement in terms of parameters such as trunk balance, fall risk, postural control abilities, functional activity and independence, which are closely related to the level of injury in patients with SCI. There is a need for a comprehensive evaluation of the patient in terms of trunk control and trunk balance, especially after a SCI defined in the thoracic segment of the medulla spinalis. In this study, male and female individuals between the ages of 18-65 years with SCI with thoracic level involvement who continue their routine treatment at the Neurological Rehabilitation Unit of Afyonkarahisar University of Health Sciences Health Application Center Department of Physical Therapy and Rehabilitation will be included. The aim of the study is to examine the relationship between trunk balance, trunk position sense, wheelchair skills and functional independence status of the participants. The findings to be obtained after the study will be analyzed in patients with SCI at the thoracic level.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with traumatic or nontraumatic spinal cord injury,
* Having a thoracic injury level (T1-T12),
* At least 6 months have passed since the SKY injury,
* To have 90 degrees of shoulder flexion and abduction in both upper extremities,
* Be over 18 years of age,
* To be able to sit in a wheelchair without support and use a manual wheelchair independently,
* Volunteering to participate in the study.

Exclusion Criteria:

* Having a systemic disease,
* Report a diagnosis of cardiovascular disease,
* Report musculoskeletal pain or pathology involving the upper extremity,
* Patients with intracardiac defibrillators,
* Presence of open wound.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with spinal cord injury who are being treated in the Department of Physical Therapy and Rehabilitation at Afyonkarahisar University of Health Sciences Health Application Center and who have thoracic level involvement and can use a manual wheelchair independently.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Modified Functional Reach Test | Baseline
  The Modified Functional Reach Test (MFRT) is an assessment tool designed to measure an individual's stability and balance by evaluating their ability to reach forward while maintaining a standing position. It involves asking the participant to extend their arm forward as far as possible without moving their feet, with the distance recorded in centimeters. This test helps identify fall risk and assess functional balance, particularly in older adults and individuals with balance impairments.
T-shirt Test | Baseline
  The T-shirt Test is a functional assessment used to evaluate the upper body mobility and coordination of individuals, particularly those with spinal cord injuries or other disabilities. During the test, participants are asked to put on and take off a T-shirt while seated in a wheelchair, which assesses their ability to perform daily activities. It measures aspects such as trunk control, upper limb function, and overall independence, providing insights into the participant's ability to manage clothing tasks in real-life situations.
The Trunk Control Test | Baseline
  The Trunk Control Test (TCT) is an assessment tool used to evaluate trunk stability and control in individuals with spinal cord injury (SCI). It involves tasks that assess the ability to maintain balance while seated and perform movements such as reaching, twisting, and turning. The test typically includes three components: static sitting balance, dynamic reaching, and trunk rotation.

SECONDARY OUTCOMES:
Trunk position sense | Baseline
  A digital inclinometer (Baseline Digital Inclinometer) will be used during the measurements. Each participant will be given a practice trial and the measurement will be repeated 3 times after the completion of the practice trial. The test procedure will be performed with the inclinometer fixed at the level of the T4 spinal process followed by active trunk flexion at a 30 degree angle. The participant will be asked to maintain and memorize this position for 5 seconds with eyes open. The participant will then be placed in a neutral position and instructed to repeat the target position with closed eyes as accurately as possible. The patient will be asked to verbally report that they have reached the same position. The absolute values of the difference between the angle values in the position taken by the patient and the 30-degree value will be recorded. Body Reposition Error will be recorded by averaging a total of 3 trials
The Wheelchair Skills Test | Baseline
  The Wheelchair Skills Test (WST) is an assessment designed to evaluate an individualls proficiency in using a wheelchair. It involves a series of tasks that simulate real-life scenarios, such as maneuvering in tight spaces, ascending and descending ramps, and navigating various surfaces.
The Spinal Cord Independence Measure | Baseline
  The Spinal Cord Independence Measure (SCIM III) is a comprehensive tool used to assess functional independence in individuals with spinal cord injuries. It evaluates three main domains: self-care, respiration and sphincter management, and mobility.

OTHER OUTCOMES:
Frequency of falls | Baseline
  Participants will be asked to retrospectively report the number of falls that have occurred in the previous six months and the amount of previous training they have received in fall prevention and transfer skills. Using the World Health Organization definition, a fall is defined as "an unintentional fall to the ground, floor or other lower level, excluding an intentional change of position to rest against furniture, walls or other objects"

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No